CLINICAL TRIAL: NCT06450470
Title: Multicenter, Randomized Study Evaluating the Use of a Non-sutured Sterile Freeze-dried Amniotic Membrane Post Crosslinking in Subjects With Progressive Keratoconus
Brief Title: Use of a Freeze-dried Amniotic Membrane Post Crosslinking in Subjects With Progressive Keratoconus
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GMALC; 2024-A00004-43 (Registry Identifier: IDRCB)
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Progressive Keratoconus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic lens alone (Active Comparator)
  Interventions: Device: Therapeutic lens alone
- Therapeutic lens + amniotic membrane (Visio-AMTRIX) (Experimental)
  Interventions: Combination Product: Therapeutic lens + amniotic membrane (Visio-AMTRIX)

INTERVENTIONS:
Device: Therapeutic lens alone — Therapeutic lens will be apposed on the patient's eye after crosslinking. Therapeutic lens will be maintained without interruption until the first postoperative visit (Day 2) when it will be removed by the investigator.
  Arms: Therapeutic lens alone
Combination Product: Therapeutic lens + amniotic membrane (Visio-AMTRIX) — Amniotic membrane (Visio-AMTRIX) will be apposed under therapeutic lens on the patient's eye after crosslinking. Amniotic membrane and therapeutic lens will be maintained without interruption until the first postoperative visit (Day 2) when it will be removed by the investigator.
  Arms: Therapeutic lens + amniotic membrane (Visio-AMTRIX)

SUMMARY:
Crosslinking is a therapeutic technique used to increase the rigidity of the cornea in order to slow or stop progression of keratoconus. The main complication of the treatment of keratoconus by crosslinking is postoperative pain due to the removal of the corneal epithelium. Currently, the management of pain is done through the administration of artificial tears and paracetamol. The amniotic membrane is a biological tissue used in ophthalmology to treat injuries of the surface of the eye. It has healing and analgesic properties.

The objective of this multicenter randomized study is to evaluate the benefit of placing an amniotic membrane on the eye post-crosslinking to reduce pain and promote corneal healing.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between 18 and 65 years old.
* Indication for accelerated conventional crosslinking.
* Patient with progressive keratoconus (increase in Kmax of ≥ 0.5 diopters in 3 to 6 months or ≥ 1 diopter in 3 to 12 months with loss of 10 microns on minimum pachymetry in 3 to 12 month).
* Patient suffering from keratoconus with a compatible topographic form (Kmax ≥ 47.0 diopters (D) and difference inferior-superior of 1.5 D).
* Patient with a minimum corneal thickness greater than 400 microns.
* Informed and consenting patient.
* Patient physically and mentally capable of completing the post-operative pain assessment self-questionnaire.
* Patient having signed the informed consent of the French Ophthalmology Society for crosslinking.
* Patient affiliated to a social security system or beneficiary of such a system.

Exclusion Criteria:

* Woman without effective means of contraception, pregnant or breastfeeding.
* Patient who has already benefited from a crosslinking procedure on one of the eyes.
* Patient with a history of refractive surgery on one of the eyes.
* Patient with an intracorneal ring segment on one of the eyes.
* Patient suffering from a serious systemic pathology (autoimmune and/or immunodepressive)
* Patient with a psychiatric pathology.
* Patient on long-term analgesics and/or corticosteroids.
* Indication of crosslinking outside the classic protocol.
* Patient with central corneal opacity.
* Patient suffering from a severe dry eye syndrome or a neurotrophic keratitis.
* Patient with a history of ocular herpes.
* Patient with a history of ocular varicella-zoster virus infection.
* Patient with glaucoma.
* Patient treated with topical cyclosporine in the last 6 months.
* Patient deprived of liberty by a judicial or administrative decision.
* Patient subject to a legal protection measure or unable to express their consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Difference between the level of ocular pain experienced by patients treated with therapeutic lens + amniotic membrane (experimental) and by patients treated with therapeutic lens alone (active comparator) | Day 0 bedtime, Day 1 wake-up, Day 1 bedtime, Day 2 wake-up, Day 2 consultation
  Pain evaluated from 0: no pain to 10: worst imaginable pain on visual analog scale (VAS)
Difference in analgesic consumption between patients treated with a therapeutic lens + amniotic membrane (experimental) and patients treated with a therapeutic lens alone (active comparator) | Day 0, Day 1, Day 2
  Amount in grams of analgesic consumed per day

SECONDARY OUTCOMES:
Difference in visual acuity between eyes treated with therapeutic lens + amniotic membrane (experimental) and eyes treated with therapeutic lens alone (active comparator) | Week 6
  Determination of logMAR values of best corrected visual acuity
Difference in corneal cicatrisation between eyes treated with therapeutic lens + amniotic membrane (experimental) and eyes treated with therapeutic lens alone (active comparator) | Day 2, (Day 7), Week 6
  Healing evaluated under slit lamp by fluorescein examination
Difference in corneal thickness between eyes treated with therapeutic lens + amniotic membrane (experimental) and eyes treated with therapeutic lens alone (active comparator) | Week 6
  Corneal thickness evaluated by anterior segment optical coherence tomography.
Difference in topographic parameters (Kmax, inferior-superior) between eyes treated with therapeutic lens + amniotic membrane (experimental) and eyes treated with therapeutic lens alone (active comparator) | Week 6
  Topographic parameters (Kmax, inferior-superior) evaluated by corneal topography
Difference in dryness between eyes treated with therapeutic lens + amniotic membrane (experimental) and eyes treated with therapeutic lens alone (active comparator) | Week 6
  Dry eye and effect on vision evaluated between 0 (no disability) and 100 (greater disability) using Ocular Surface Disease Index (OSDI)

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU de Brest, Brest
  - Hospices Civils de Lyon, Lyon
  - Assistance Publique - Hôpitaux de Marseille, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - Hôpital National de la Vision des Quinze-Vingts, Paris
  - CHU de Saint-Etienne, Saint-Priest-en-Jarez
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No